CLINICAL TRIAL: NCT05672199
Title: A Phase 2 Long-Term Extension (LTE) Study to Evaluate The Safety and Efficacy of Efavaleukin Alfa in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Long-term Safety and Efficacy of Efavaleukin Alfa in Participants With Moderately to Severely Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The parent study 20170104 was terminated due to the study meeting a prespecified futility rule. Consequently, this study was terminated.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210210; 2022-001686-12 (EudraCT Number)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; UC; Moderately to severely active ulcerative colitis; Efavaleukin alfa; AMG 592
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants who were receiving the placebo during the dose-finding study (study 20170104) that decided to continue onto this long-term extension study will continue to receive the placebo.
  Interventions: Drug: Placebo
- Efavaleukin Alfa Dose 1 (Low Dose) (Experimental): Participants who were receiving efavaleukin alfa dose 1 during the dose-finding study (study 20170104) that decided to continue onto this long-term extension study will continue to receive efavaleukin alfa dose 1.
  Interventions: Drug: Efavaleukin alfa
- Efavaleukin Alfa Dose 2 (Moderate Dose) (Experimental): Participants who were receiving efavaleukin alfa dose 2 during the dose-finding study (study 20170104) that decided to continue onto this long-term extension study will continue to receive efavaleukin alfa dose 2.
  Interventions: Drug: Efavaleukin alfa
- Efavaleukin Alfa Dose 3 (High Dose) (Experimental): Participants who were receiving efavaleukin alfa dose 3 during the dose-finding study (study 20170104) that decided to continue onto this long-term extension study will continue to receive efavaleukin alfa dose 3.
  Interventions: Drug: Efavaleukin alfa

INTERVENTIONS:
Drug: Efavaleukin alfa — Subcutaneous (SC) injection
  Other Names: AMG 592
  Arms: Efavaleukin Alfa Dose 1 (Low Dose); Efavaleukin Alfa Dose 2 (Moderate Dose); Efavaleukin Alfa Dose 3 (High Dose)
Drug: Placebo — SC injection
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the long-term safety and tolerability of efavaleukin alfa in participants with moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Participant has completed the week 52 endoscopy in the phase 2 dose-finding parent study (20170104) and who in the opinion of the investigator may benefit from continued treatment.

Exclusion criteria:

* Permanent discontinuation of investigational product during the 52- week phase 2 dose finding parent study (20170104) for any reason
* Female subjects of reproductive potential must agree not to donate eggs during the study and for 6 weeks after receiving the last dose of investigational product.

Disease Related:

* Adenoma and dysplasia exclusion criteria:

  * Any current sporadic adenoma without dysplasia (adenomatous polyps occurring proximal to known areas of colitis) that has not been removed.
  * Dysplasia occurring in flat mucosa, sporadic adenomas containing dysplasia, and dysplasia-associated lesions or masses will be managed as follows:
* Any history or current evidence of high-grade dysplasia.
* Any history or current evidence of dysplasia occurring in flat mucosa.
* This includes histopathology reporting indefinite for dysplasia, low-grade dysplasia, and high-grade dysplasia.
* Any history or current evidence of a nonadenoma like dysplasia associated lesions or masses, with or without evidence of dysplasia.
* Any current sporadic adenoma containing dysplasia or any current adenoma-like dysplasia-associated lesions or masses that has not been removed.

Other Medical Conditions:

* Any malignancy diagnosed during parent Study 20170104, including evidence of cutaneous basal or squamous cell carcinoma or melanoma
* Active infection (including chronic, acute, recurrent, opportunistic infections) at the time of eligibility evaluation requiring intravenous (IV) anti-infectives or hospitalization (infections requiring oral and/or topical anti-infective[s] for > 7 days may be allowed in consultation with the Amgen physician).
* Required systemic corticosteroid use for any indication other than ulcerative colitis. The only exception is corticosteroids used for the treatment of adrenal insufficiency are allowed.
* Plan to receive a live (attenuated) vaccine during the treatment period and up to 6 weeks after the last dose of investigational product in the long term extension study.

Prior/Concurrent Clinical Study Experience:

* Currently receiving treatment in another investigational device or drug study. Other investigational procedures while participating in this study are excluded.

Other Exclusions:

* Female participants who are pregnant or breastfeeding or planning to become pregnant or breastfeed during study and for an additional 6 weeks after the last dose of investigational product.
* Female participants of childbearing potential unwilling to use protocol specified method of contraception see Appendix 5 (Section 11.5) during treatment and for an additional 6 weeks after the last dose of investigational product.
* Participant has known sensitivity to any of the products to be administered during dosing with the exception of participants who exhibited sensitivity in parent Study 20170104 but did not result in treatment discontinuation.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (e.g., Clinical Outcome Assessments) to the best of the participant and investigator's knowledge.
* Participant has a history or evidence of any other clinically significant disorder (including laboratory abnormalities), condition, or disease that, in the opinion of the investigator or Amgen physician, if consulted would pose a risk to participant safety, or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 to Week 110

SECONDARY OUTCOMES:
Number of Participants with Clinical Response at Week 52 | Week 52
Number of Participants with Clinical Response at Week 104 | Week 104
Number of Participants with Clinical Remission at Week 52 | Week 52
Number of Participants with Clinical Remission at Week 104 | Week 104
Number of Participants with Durable Clinical Remission at Week 52 | Week 52
Number of Participants with Durable Clinical Remission at Week 104 | Week 104
Number of Participants with Endoscopic Remission at Week 52 | Week 52
Number of Participants with Endoscopic Remission at Week 104 | Week 104
Number of Participants with Histologic Remission at Week 52 | Week 52
Number of Participants with Histologic Remission at Week 104 | Week 104
Number of Participants with Corticosteroid-free Remission | Week 52
  Measured in participants receiving corticosteroids at randomization of parent Study 20170104.
Number of Participants with Corticosteroid-free Remission | Week 104
  Measured in participants receiving corticosteroids at randomization of parent Study 20170104.
Number of Participants with Combined Endoscopic and Histologic Remission at Week 52 | Week 52
Number of Participants with Combined Endoscopic and Histologic Remission at Week 104 | Week 104
Number of Participants with Symptomatic Remission at Week 52 | Week 52
Number of Participants with Symptomatic Remission at Week 104 | Week 104
Change from Baseline of Study 20170104 in Histological Score (Geboes) at Week 52 | Baseline of Study 20170104 to Week 52 of Long Term Extension Study (up to approximately 104 weeks)
Change from Baseline of Study 20170104 in Histological Score (Geboes) at Week 104 | Baseline of Study 20170104 to Week 104 of Long Term Extension Study (up to approximately 156 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (25):
- United States (3):
  - Santa Maria Gastroenterology Medical Group, Santa Maria, California
  - Indian Health Service Health Research, Kissimmee, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
- Argentina (3):
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Clinica Independencia, Munro, Buenos Aires
  - Cer Instituto Medico, Quilmes, Buenos Aires
- Diagnostic-Consultative Center Convex EOOD, Sofia, Bulgaria
- Herlev Hospital, Herlev, Denmark
- Universitaetsklinikum Ulm, Ulm, Germany
- Hungary (3):
  - MIND Klinika Kft, Budapest
  - Clinexpert Kft, Budapest
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Japan (3):
  - Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Ome Medical Center, Ome-shi, Tokyo
- Clinica de Investigacion en Reumatologia y Obesidad SC, Guadalajra, Jalisco, Mexico
- Poland (2):
  - NZOZ Twoje Zdrowie EL Spzoo, Elblag
  - Centrum Medyczne Melita Medical, Wroclaw-Krzyki
- Romania (3):
  - Clinica Medicum, Bucharest
  - Memorial Healthcare International SRL, Bucharest
  - Spitalul Clinic Colentina, Bucharest
- Wonju Severance Christian Hospital, Wonju-si, Gangwon-do, South Korea
- Intesto BE, Bern, Switzerland
- Turkey (Türkiye) (2):
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com